CLINICAL TRIAL: NCT03314584
Title: Long Term Efficacy of rTMS in Managing MTBI-related Headache
Brief Title: Managing Mild Traumatic Brain Injury Related Headaches With Repetitive Transcranial Magnetic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2506-I; H170053 (Other: VA San Diego Healthcare System)
Record Dates: First submitted 2017-10-04; First posted 2017-10-19 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Traumatic Brain Injury (TBI)
Keywords: TBI; traumatic brain injury; transcranial magnetic stimulation; headache
MeSH Terms: conditions — Brain Injuries, Traumatic; Headache | interventions — Transcranial Magnetic Stimulation; Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blinded study where only the statistician is aware of the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcranial Magnetic Stimulation (Experimental): Active-repetitive transcranial magnetic stimulation (rTMS) at the left motor cortex.
  Interventions: Device: Transcranial Magnetic Stimulation; Diagnostic Test: Magnetic resonance imaging (MRI)
- Sham Transcranial Magnetic Stimulation (Sham Comparator): Sham rTMS will consist of the same parameters as active, however, the subject will not receive the actual magnetic stimulation to the left motor cortex.
  Interventions: Device: Sham Transcranial Magnetic Stimulation; Diagnostic Test: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Active-repetitive transcranial magnetic stimulation (rTMS) at the left motor cortex.
  Arms: Transcranial Magnetic Stimulation
Device: Sham Transcranial Magnetic Stimulation — Sham rTMS will consist of the same parameters as active, however, the subject will not receive the actual magnetic stimulation to the left motor cortex due to the use of a double sided Active/Sham coil used specifically for research studies.
  Arms: Sham Transcranial Magnetic Stimulation
Diagnostic Test: Magnetic resonance imaging (MRI) — Brain imaging will be done via MRI prior to the first rTMS/Sham TMS session. Imaging will allow investigators to target specific areas in the brain.

SUMMARY:
Persistent headache is one of the most common debilitating symptoms in military personnel suffering from mild traumatic brain injury (MTBI). This study aims to assess the long-term effect of repetitive transcranial magnetic stimulation (rTMS) in managing MTBI related headaches for up to 2-3 months by comparing the treatment effect of active-rTMS to sham-rTMS.

DETAILED DESCRIPTION:
Headache is one of the most common debilitating chronic pain conditions in either active or retired military personnel with MTBI. This high prevalence of persistent chronic headache is often associated with neuropsychological dysfunction in mood, attention, and memory, which casts a profound negative impact on patients' quality of life and increases stress in their caregivers. Unfortunately, as witnessed by the investigators in their clinical practices, conventional pharmacological treatments for MTBI related headache (MTBI-HA) has not been shown to be effective and drugs such as narcotics contain many long-term untoward psychosomatic and abusive side effects. This calls for an urgent need in developing alternate and innovative long-term headache management strategies for this rapidly increasing patient population.

Coinciding with other published treatment protocols related to traumatic brain injury and pain, this initial clinical evidence provides compelling support for the current proposal aiming to assess the effect of a longer duration of rTMS protocol in managing MTBI-HA for up to 10 weeks after the initiation of the treatment. Given existing treatment options for MTBI-HA are limited, validating such a non-pharmacological and non-invasive treatment option will significantly enhance the capability of the VA healthcare system in caring for this rapidly increasing patient population.

1. PRE-TREATMENT PHASE (weeks 1-2) consists of Visit 1 (Screening Visit) and Visit 2 (Pre-treatment Assessments);
2. TREAMENT PHASE (week 3-4) consists of Visits 3-12 (Neuronavigation guided rTMS consisting of 10 weekday treatments at >24 and < 72 hours apart, weekends excluded, maximum 5 weeks for treatment completion) rTMS will take place in Building 23 Room 105 at the VASDHS; and
3. POST-TREATMENT PHASE (week 5-14) consists of two initial weekly visits (Visits 13&14) and two additional biweekly visits (Visits 15&16) and one monthly visit (Visit 17).

Brain anatomical and functional MRI will be performed within 72 hours after Visits 2 and 13. Subjects will be required to fill out headache diary between assessment visits. Headache assessments along with quality of life, mood and functions assessments will be carried out at Visits 1,2, and 13--17. This frequency of treatment and duration of follow-up is in line with recently published rTMS articles related to TBI, headache and pain, and also in accordance with the 3-month post treatment initiation follow-up guideline/recommendation.

ELIGIBILITY:
Inclusion Criteria:

* The following diagnostic criteria for MTBI based on the 1993 American Congress of Rehabilitation Medicine and recent recommendation from the DOD, and the current diagnostic criteria adopted by the VASDHS TBI Clinic will be used for the study. A traumatically induced physiological disruption of brain function, as manifested by at least one of the following:
* any loss of consciousness
* any loss of memory for events immediately before or after the accident
* any alteration in mental state at the time of the accident, e.g.:

  * feeling dazed
  * disoriented
  * confused)
* Focal neurologic deficit (s) that may or may not be transient but where the severity of the injury does not exceed the following:

  * loss of consciousness of approximately 30 min or less
  * after 30 min, an initial Glasgow Coma Scale score of 13-15
  * post-traumatic amnesia not greater than 24 hrs
* In addition, the following established diagnostic criteria for " Persistent headache attributed to mild traumatic injury headache" based on the International Classification of Headache Disorder (ICHD-3) will be applied to the study subjects:

  * A. Any headache fulfilling criteria C and D
  * B. Traumatic injury to the head has occurred
  * C. Headache is reported to have developed within 7 d after one of the following:
  * 1. injury to the head
  * 2. regaining of consciousness following the injury
  * 3. discontinuation of medication(s) that impairs the ability to sense or report headache following the injury
  * D. Headache persists for >3 mo after injury to the head
  * E. Not better accounted for by another ICHD-3 diagnosis

Additional Inclusion Criteria:

* no prior experience of TMS treatment
* average persistent headache intensity more than 30 on the 0-100 mechanical visual analog scale(M-VAS) at the screening visit (visit 1) and average persistent headache intensity score greater than 3/10 on a numerical rating scale (NRS) reported in the headache diary (between visits 1&2)
* no history of daily persistent headache prior to the MTBI incidence

Exclusion Criteria:

* pregnancy; To be eligible for the study and to ensure no pregnancy risk, you will need to utilize contraception or practice abstinence until your study participation is completed
* history of pacemaker implant
* any ferromagnetic material in the brain or body that would prohibit the patients from having a brain MRI, e.g.:

  * bullet fragment
  * shrapnel
  * device implant
* history of dementia, major psychiatric or life threatening diseases
* presence of any other chronic neuropathic pain states;
* history of seizure
* pending litigation
* lack of ability to understand the experimental protocol and to adequately communicate in English
* history of chronic headache diagnoses such migraine, tension or cluster headaches prior to the incidence of MTBI.
* history of chronic headache prior to the MTBI incidence at a frequency more than once a month lasting more than one hour.
* evidence in the chart of recent exacerbation of depressive or anxiety symptoms, active substance dependence, suicidal intent or attempt within the previous month, and/or current psychotic symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yick Leung, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leung A, Ho M, Vaninetti M, Krug P, Rutledge T, Lin L, Tsai A, Le L, Rimmele C, Lee R, Golshan S. Long-term Efficacy of Repetitive Transcranial Magnetic Stimulation at Motor Cortex for Mild Traumatic Brain Injury-Related Headaches. Neuromodulation. 2025 Oct 18:S1094-7159(25)01033-5. doi: 10.1016/j.neurom.2025.09.308. Online ahead of print. PMID 41109991

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Started (Does not include subjects who enrolled in the study but withdrew before receiving a group and study interventions.) | 38 | 41
Completed | 31 | 38
Not Completed | 7 | 3
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 4 | 0

BASELINE CHARACTERISTICS:
Population: Subjects were included if they completed up to at least their 1-month follow up assessment visit (visit 16). Some subjects were included that were missing some of their visit 14-16 data but had data past that point (visits 17 and 18). This was done to allow for ample post-intervention data for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation | Total
Number analyzed (Participants) | 32 | 38 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.88 (11.07) | 40.76 (7.76) | 39.44 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 26 | 32 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 24 | 28 | 52
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 4 | 5 | 9
  White | 23 | 23 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 38 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Headache Days Per Week
Description: The outcome measure will be quantified through the headache diary log that tracks the intensity, frequency and duration of MTBI-headaches (MTBI-HA). Baseline data includes all logs from the start of the study until the start of treatment. Post-intervention data looked at the time between the 3-month follow-up and the previous visit.
Time Frame: The measure will be assessed daily from baseline to the 3-month post-treatment follow up (treatment occurred for 2-5 weeks starting in week 3).
Population: Some subjects are missing their 3-month follow up data due to it not being collected.
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 32 | 38
days/week
  Pre-intervention persistent headache frequency | 4.2 (2.9) | 4.6 (2.0)
  Post-intervention (3-months after TX) persistent headache frequency: number analyzed (Participants) | 30 | 38
  Post-intervention (3-months after TX) persistent headache frequency | 3.1 (2.3) | 4.3 (1.9)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Superiority; p < 0.000, Mixed Models Analysis; F=21.662, df = 1

2. Primary Outcome: Number of Days With Debilitating MTBI-headaches Per Week.
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Some subjects were excluded from the pre-intervention or post-intervention data due to missing data. Subjects did not need both to be included in the analysis. The number analyzed below reflects that total subjects with valid data for that group and time point.
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 30 | 38
days/week
  Pre-intervention debilitating headache frequency | 2.1 (2.0) | 2.1 (1.9)
  Post-intervention (3-months after TX) debilitating headache frequency | 1.3 (1.8) | 1.8 (1.7)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Superiority; p = 0.004, Mixed Models Analysis; F=5.624, df=1

3. Primary Outcome: Duration of Debilitating MTBI-headaches (Hours).
Description: as for outcome 1
Time Frame: The measure will be assessed daily from baseline to the 3-month post-treatment follow up (treatments occurred for 2-5 weeks starting in week 3).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 30 | 38
hours
  Pre-intervention debilitating headache duration | 3.5 (1.6) | 5.5 (4.6)
  Post-intervention (3-months after TX) debilitating headache duration | 4.3 (3.3) | 5.0 (4.3)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Superiority; p = 0.046, Mixed Models Analysis; F=3.092, df=1

4. Primary Outcome: Average Interference (0-10) of Headaches in Daily Activities.
Description: The outcome measure will be quantified through the headache diary log that tracks the intensity, frequency, duration, and interference of MTBI-headaches (MTBI-HA). A score of 0 for interference would indicate no interference in daily activities while a score of 10 would indicate complete interference (e.g. the subject could not get out of bed and go to work due to their pain). Baseline data includes all logs from the start of the study until the start of treatment. Post-intervention data looked at the time between the 3-month follow-up and the previous visit.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 30 | 38
score on a scale
  Pre-intervention debilitating headache interference | 6.9 (1.5) | 6.6 (1.8)
  Post-intervention (3-months after TX) debilitating headache interference | 5.8 (2.1) | 5.7 (2.6)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Superiority; p = 0.018, Mixed Models Analysis; F=4.022, df=1

5. Primary Outcome: Baseline vs Post-Treatment HIT-6 Scores (36-78).
Description: The outcome measure is measuring headache impact on quality of life and will be quantified through the self-assessed Headache Impact Test (HIT-6). Each question ranges from 6-13 and the total score ranges from 36 to 78. The assessment indicates the effect that headaches have on normal daily life and ability to function with a higher score indicating more interference in daily life and function.
Time Frame: The measure will be assessed every visit from baseline to the 3-month post-treatment follow up (treatment occurred for 2-5 weeks starting in week 3).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 32 | 38
score on a scale
  Pre-intervention HIT-6 total score.: number analyzed (Participants) | 32 | 37
  Pre-intervention HIT-6 total score. | 65.2 (4.8) | 65.1 (6.5)
  Post-intervention (3-months post TX) HIT-6 total score.: number analyzed (Participants) | 28 | 38
  Post-intervention (3-months post TX) HIT-6 total score. | 60.7 (8.8) | 60.3 (8.8)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Superiority; p = 0.598, Mixed Models Analysis; F=0.279, df=1

6. Primary Outcome: Change From Baseline to Post-Treatment HDRS-17 Scores
Description: The outcome measure will be measuring depression scores and will be quantified through the administered Hamilton Scale for Depression. This contains 17 items to be rated (HDRS-17), but four other questions are not added to the total score and are used to provide additional clinical information. Each item on the questionnaire is scored on a 3 or 5 point scale, depending on the item, and the total score is compared to the corresponding descriptor. The total score ranges from 0 to 53 and is calculated from adding together the first 17 questions. A higher score indicated more severe depression.
Time Frame: The measure will be assessed each visit from baseline to the 3-month post-treatment follow up (treatment occurred for 2-5 weeks starting in week 3).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 33 | 38
score on a scale
  Pre-intervention HRSD total score.: number analyzed (Participants) | 33 | 37
  Pre-intervention HRSD total score. | 14.5 (7.4) | 16.5 (7.1)
  Post-intervention (3-months post TX) HRSD total score. | 11.8 (8.8) | 12.3 (7.8)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Superiority; p = 0.296, Mixed Models Analysis; F=1.101, df=1

7. Primary Outcome: Connors Continuous Performance Test Score.
Description: The outcome measure quantified through the Connors continuous performance test will be sustained and selective attention. This is administered on a laptop and is automatically scored. Key performance indicators are reported as T-scores (mean of 50, SD = 10) and percentiles. T-scores are compared to the normative sample. Variability measure which looked at response speed consistency and indicated fluctuations in attention. A higher score indicated more fluctuations.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 26 | 32
T-Score
  Pre-intervention CPT-3 Variability score. | 58.0 (15.2) | 66.1 (19.0)
  Post-intervention (3-months post TX) CPT-3 Variability score.: number analyzed (Participants) | 18 | 26
  Post-intervention (3-months post TX) CPT-3 Variability score. | 61.3 (18.8) | 56.1 (12.9)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Superiority; p = 0.033, Mixed Models Analysis; F=4.672, df = 1

8. Primary Outcome: Brief Pain Inventory Global Score.
Description: The outcome will measure global pain through the brief pain inventory assessment. Pain will be recorded at it's worst, it's best and on average over the previous 24 hours on a 0 to 10 scale These scores are reflected in questions 3-6 of the assessment and will be averaged together to give an overall average pain level score with a higher value reflecting more pain. Then the pain's impact on general activity, mood, walking ability, normal work, relationships, sleep and enjoyment of life will be measured on a 0 to 10 scale and averaged for an overall pain score. These scores are reflected in question 9a-g and will be averaged together to give an overall average pain interference level with a higher value indicating more interference in daily life.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 25 | 33
score on a scale
  Pre-intervention BPI overall score.: number analyzed (Participants) | 25 | 30
  Pre-intervention BPI overall score. | 5.1 (1.4) | 5.5 (1.8)
  Post-intervention (3-months post TX) BPI overall score.: number analyzed (Participants) | 23 | 33
  Post-intervention (3-months post TX) BPI overall score. | 4.2 (2.6) | 4.3 (2.4)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Superiority; p = 0.606, Mixed Models Analysis; F=0.268, df=1

9. Primary Outcome: Hopkins Verbal Learning Test (HVLT-R) Total Scores
Description: The Hopkins Verbal Learning Test (HVLT-R) will be used to measure memory. In this assessment, 12 words are taught and subjects are tasked to recall those words in three difference trials. When scoring the HVLT-R, the number of words recalled are summed to calculate a total recall score which ranges from 0-36 with higher values indicating more words being recalled.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 33 | 38
score on a scale
  Pre-intervention HVLT-R total recall score. | 23.5 (4.6) | 21.9 (5.4)
  Post-intervention (3-months post TX) HVLT-R total recall score.: number analyzed (Participants) | 31 | 38
  Post-intervention (3-months post TX) HVLT-R total recall score. | 24.2 (5.8) | 23.7 (6.7)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Superiority; p = 0.287, Mixed Models Analysis; F=1.142, df=1

10. Primary Outcome: Stroop Test Score
Description: The Stroop test was administered to assess cognitive functioning performance. In the test, the participant must demonstrate inhibition of cognitive interference by naming the color of the colored word instead of the word itself based on the observation that normal individuals can read words much faster than they can identify and name colors. This follows two other trials where the participant just reads the words aloud and another trial of the participant just identifying the color of a series of x's. Each trial, the participant was given 45 second to identify as many colors as they could. There is no maximum score for this assessment. This assessment is scored by the number of items they were able to correctly read out rather than on a T-score. A higher score indicated higher cognitive functioning.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of words
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 27 | 31
Number of words
  Pre-intervention Stroop color word total score. | 36.6 (13.0) | 37.2 (14.2)
  Post-intervention (3-months post TX) Stroop color word total score.: number analyzed (Participants) | 23 | 29
  Post-intervention (3-months post TX) Stroop color word total score. | 44.2 (12.2) | 43.6 (9.5)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Superiority; p = 0.049, Mixed Models Analysis; F=4.039, df=1

11. Primary Outcome: Average Intensity of Persistent Headaches.
Description: The outcome measure will be quantified through the headache diary log that tracks the intensity, frequency and duration of MTBI-headaches (MTBI-HA). Intensity was rated on a scale of 0-10 with 0 indicating no pain and 10 indicating the worst pain they have experienced. Baseline data includes all logs from the start of the study until the start of treatment. Post-intervention data looked at the time between the 3-month follow-up and the previous visit.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 32 | 38
score on a scale
  Pre-intervention persistent headache intensity | 5.0 (1.3) | 4.7 (1.5)
  Post-intervention (3-months after TX) persistent headache Intensity | 3.8 (1.5) | 3.9 (1.7)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Superiority; p = 0.338, Mixed Models Analysis; F=1.084, df=1

12. Primary Outcome: Average Intensity of Debilitating Headaches.
Description: The outcome measure will be quantified through the headache diary log that tracks the intensity, frequency and duration of MTBI-headaches (MTBI-HA). Intensity was rated on a scale of 0-10 with 0 indicating no pain and 10 indicating the worst pain they have experience. Baseline data includes all logs from the start of the study until the start of treatment. Post-intervention data looked at the time between the 3-month follow-up and the previous visit.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 32 | 38
score on a scale
  Pre-intervention debilitating headache intensity | 6.6 (1.6) | 6.5 (1.7)
  Post-intervention (3-months after TX) debilitating headache Intensity | 5.8 (2.0) | 5.7 (2.4)

13. Secondary Outcome: Significant T-Values for Connectivity Between Regions.
Description: Resting state functional magnetic imaging scans and subsequent processing using CONN Toolbox were used to determine T-values. ROIs (region of interest) where determined and compared to other ROIs to assess connectivity between regions. Value of "0" indicated no significant connectivity between regions (p<0.01). The sign of the value indicated directionality of connectivity. Larger absolute values of the T-value indicated stronger connectivity.
Time Frame: Subjects will have 2 functional magnetic imaging scans, at baseline and then at the 1-week post treatment follow-up.
Population: Some subjects were excluded due to not having a resting state MRI scan performed.
Measure: Number; unit: T-value
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 28 | 35
T-value
  Left Motor Cortex (BA4) to Cingulate (BA24-31) | 4.06 | 6.12
  Left Motor Cortex (BA4) to Premotor (BA6) | 8.77 | 8.76
  Left Motor Cortex (BA4) to Premotor (BA46) | -3.23 | -3.61
  Left Motor Cortex (BA4) to Insula (BA13) | 6.57 | 5.50
  Left Motor Cortex (BA4) to Somatosensory (BA7) | 2.85 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/38 | 2/41
Other Adverse Events (participants affected / at risk) | 0/38 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial Magnetic Stimulation (N=38) | Sham Transcranial Magnetic Stimulation (N=41)
Vasovagal Response during study intervention (General disorders) | 0 (0) | 1 (1) — A transient vasovagal response occurred during the study intervention. The session was aborted and the subject was determined to be okay after a neurological exam. Subject continued the study with vital sign monitoring with no issues.
Increased sensitivity to light w/ nausea (General disorders) | 1 (1) | 0 (0) — Transient increase in light sensitivity accompanied with nausea impaired subject's ability to drive. Subject advised to wait 15 minutes after receiving intervention.
Breast Cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Subject diagnosed with breast cancer during their participation in the study (not related to study intervention).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT03314584/Prot_SAP_000.pdf